CLINICAL TRIAL: NCT05631977
Title: Prospective Acquisition of Cardiac Ultrasound Images at the Point of Care
Acronym: POCUS_ACQ
Status: Completed | Type: Observational
Sponsor: Aisap LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: POC1
Record Dates: First submitted 2022-11-17; First posted 2022-11-30 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Diagnosis
Keywords: Point of care ultrasound; Echocardiography
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- POCUS acquisition: Prospective noninterventional single arm study collection of cardiac POCUS examination according to prespecified acquisition protocol.
  Alongside POCUS images the study will also collect demographic and clinical information from the study participants and some information from the healthcare personal performing the POCUS exam (experience in US image acquisition, physician specialty or sonographer).
  Patient management will not be impacted, and usual care will follow the regular practices at the study site.
  Interventions: Other: Point of care ultrasound cardiac examination

INTERVENTIONS:
Other: Point of care ultrasound cardiac examination — The study intervention consists of a POCUS cardiac examination by site approved personal using an FDA cleared US scanner. Usual care of study participants will not be impacted.

SUMMARY:
The present study is a preparatory step towards a multi-reader multi case (MRMC) randomized fully crossed study. As POCUS images are frequently not stored and not methodically acquired using a standardized image acquisition protocol this study will collect cardiac POCUS images in a prespecified manner.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 21 or more

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Unstable clinical condition according to PI clinical judgment
2. Presence of prosthetic cardiac valve at any position and any type
3. Pregnancy or lactation
4. Contact isolation due to infections disease
5. Presence of left ventricular assist device (LVAD)
6. Know existence of congenital heart disease
7. Prosthetic cardiac valve, any
8. BMI 40 or greater
9. Clinical conditions that do not permit a POCUS study according to the judgment of the investigators or treating physicians
10. History of lung resection
11. Known poor cardiac US image quality based on prior echo exams
12. Mechanical ventilation, or other situations where the required ultrasound views cannot be adequately obtained
13. Clinical instability or critical subject condition or any condition the study PI judges that the POCUS exam could adversely affect the participant

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals under the care of the cardiology institutes of the participating sites, both inpatients and outpatient clinics and services.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
POCUS QUALITY | 1 month
  Primary endpoint: Percent of POCUS exams that attain the pre-specified POCUS image quality threshold (quality standard)

SECONDARY OUTCOMES:
Subgroup analysis | 1 month
  Analysis of primary endpoint (POCUS exam quality) by the prespecified subgroups of age (above or below 65), gender, BMI group (below or above 25) and US device manufacturer.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Inova Health, Fairfax, Virginia
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No